CLINICAL TRIAL: NCT02909179
Title: mCARE II: Enhancing, Integrating and Scaling mCARE and Measuring the Impact of a Mobile Health System to Support Healthy Pregnancies and Improve Newborn Survival
Brief Title: Measuring the Impact of a Mobile Health System to Support Healthy Pregnancies and Improve Newborn Survival
Acronym: mCARE-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: mPower Social Enterprises Limited (Unknown); The JiVitA Project (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00006469
Record Dates: First submitted 2016-09-19; First posted 2016-09-21 (Estimated); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: High Perinatal Mortality; High Neonatal Mortality; Low Antenatal Care Service Utilization; Low Postnatal Care Service Utilization
Keywords: Community Health Workers, mHealth, mobile phones, ANC, PNC, essential newborn care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mCARE-II (Experimental): mCARE-II supported service provision through existing community health workforce.
  Interventions: Other: mCARE-II
- Comparison (No Intervention): Standard of care, paper-based service provision through existing community health workforce.

INTERVENTIONS:
Other: mCARE-II — mCARE-II is a package of interventions that provides guided client enumeration and follow-up support to community health workers, automated workflow scheduling, risk assessment, client prioritization and stratification and client-based demand generation messaging. These features are incorporated into a platform called OpenSRP, which integrates text message reminders, scheduling, and form submissions on the server side, and displays schedules and client lists on a tablet-based application for community health workers.
  Arms: mCARE-II

SUMMARY:
The purpose of this community-based randomized controlled trial is to test whether the mCARE-II intervention package, delivered by the existing Government of Bangladesh community health workforce, will improve neonatal and perinatal survival in a rural setting in northwestern Bangladesh. mCARE-II is a digital health intervention, which incorporates automated workload scheduling, client prioritization and risk stratification, overdue service reminders and demand generation through client side reminder messaging. The intervention package focuses on the pregnancy and early postpartum period.

DETAILED DESCRIPTION:
The aim of this study is to implement and evaluate the mCARE-II intervention package using a randomized controlled trial design. This package, supported by an mHealth application, provides workflow scheduling for guided household registration, census, pregnancy surveillance, and antenatal, postnatal, and essential newborn care visit reminders. Workflow scheduling is sorted and prioritized based on assessment of basic risk. Furthermore, the system integrates client-directed reminder SMS messages and demand-side birth notifications to schedule postnatal services immediately after birth. This will be operated by the Government of Bangladesh (GoB) community health workers, called Family Welfare Assistants (FWAs), in 18 unions of one northern district of Bangladesh who will use the system to support their routine health service delivery functions. Based on lessons learned from phase I implementation under the pilot study, additional features will be added to the intervention package, including a priority sorting algorithm to identify pregnant women and newborns with known risk factors for adverse outcomes to prioritize them for scheduled visits, a birth preparedness module to help pregnant women and their families plan for safe delivery and childbirth, and targeted newborn care counseling during late antenatal encounters. These features will be built on a scalable platform compatible with national data systems and aligned with a new global standard being advocated by WHO - the Open Smart Register Platform or OpenSRP (smartregister.org).

Based on randomization to mCARE-II or control arms by FWA catchment area, participants living in each area will receive services from their FWA, either supported by OpenSRP or according to the standard of care procedures currently in place. Performance of the FWAs and the health status of enrolled women and newborns will be monitored and evaluated by a rigorous research layer supported by a cadre of research workers who will verify services received by participants to assess exposure to and interactions with FWAs and OpenSRP. This study combines a robust RCT methodology with principles of implementation science - actual government health workers using OpenSRP to support their routine work while a cadre of highly-trained research workers collects 'gold-standard' denominator data against which to measure performance. This study is an effort to rigorously evaluate the set of mCARE-II interventions on the OpenSRP platform.

ELIGIBILITY:
Inclusion Criteria:

* Married women of reproductive age living with their husbands in the JiVitA study area in Gaibandha, Bangladesh
* Consented for participation in 8 weekly pregnancy surveillance
* Self reported as being pregnant
* Infants born to eligible, enrolled women

Exclusion Criteria:

* Women who are menopausal or sterilized
* Refused to participate in 8 weekly pregnancy surveillance

Max Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 113539 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2020-12-22 (Actual)

PRIMARY OUTCOMES:
Decrease in Neonatal Mortality | Within 43 days after birth
Decrease in perinatal mortality | 22 Weeks Gestation through the first 7 days after birth

SECONDARY OUTCOMES:
Increase in postnatal care utilization | Within 7 days of delivery/child birth
Increase in essential newborn care utilization | Within 7 days of delivery/child birth
Increase in antenatal care utilization | up to 34 weeks of pregnancy
Increase in skilled birth attendance | During child birth
Increase in immediate breastfeeding | Within first hour of life
Increase in facility-based delivery | At time of delivery
Increase in skilled birth attendance | At time of delivery

CONTACTS AND LOCATIONS:
Locations (1):
- JiVitA: Maternal and Child & Nutrition Research Site, Gaibandha, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Darmstadt GL, Bhutta ZA, Cousens S, Adam T, Walker N, de Bernis L; Lancet Neonatal Survival Steering Team. Evidence-based, cost-effective interventions: how many newborn babies can we save? Lancet. 2005 Mar 12-18;365(9463):977-88. doi: 10.1016/S0140-6736(05)71088-6. PMID 15767001
- [Background] Schiffman J, Darmstadt GL, Agarwal S, Baqui AH. Community-based intervention packages for improving perinatal health in developing countries: a review of the evidence. Semin Perinatol. 2010 Dec;34(6):462-76. doi: 10.1053/j.semperi.2010.09.008. PMID 21094420
- [Background] Jones G, Steketee RW, Black RE, Bhutta ZA, Morris SS; Bellagio Child Survival Study Group. How many child deaths can we prevent this year? Lancet. 2003 Jul 5;362(9377):65-71. doi: 10.1016/S0140-6736(03)13811-1. PMID 12853204
- [Background] Baqui AH, Rosen HE, Lee AC, Applegate JA, El Arifeen S, Rahman SM, Begum N, Shah R, Darmstadt GL, Black RE. Preterm birth and neonatal mortality in a rural Bangladeshi cohort: implications for health programs. J Perinatol. 2013 Dec;33(12):977-81. doi: 10.1038/jp.2013.91. Epub 2013 Aug 15. PMID 23949837
- [Background] Jo Y, Labrique AB, Lefevre AE, Mehl G, Pfaff T, Walker N, Friberg IK. Using the lives saved tool (LiST) to model mHealth impact on neonatal survival in resource-limited settings. PLoS One. 2014 Jul 11;9(7):e102224. doi: 10.1371/journal.pone.0102224. eCollection 2014. PMID 25014008
- [Background] G Mehl, L Vasudevan, L Gonsalves, M Berg, T Seimon, M Temmerman, AB Labrique. Harnessing mHealth in low-resource settings to achieve universal access to health. In: Marsch LA, Lord SE, Dallery J, editors. Transforming Behavioral Health Care with Technology: The State of the Science. Oxford University Press; 2014
- [Background] Labrique AB, Vasudevan L, Kochi E, Fabricant R, Mehl G. mHealth innovations as health system strengthening tools: 12 common applications and a visual framework. Glob Health Sci Pract. 2013 Aug 6;1(2):160-71. doi: 10.9745/GHSP-D-13-00031. eCollection 2013 Aug. PMID 25276529
- [Background] Lund S, Hemed M, Nielsen BB, Said A, Said K, Makungu MH, Rasch V. Mobile phones as a health communication tool to improve skilled attendance at delivery in Zanzibar: a cluster-randomised controlled trial. BJOG. 2012 Sep;119(10):1256-64. doi: 10.1111/j.1471-0528.2012.03413.x. Epub 2012 Jul 17. PMID 22805598
- [Background] Tran MC, Labrique AB, Mehra S, Ali H, Shaikh S, Mitra M, Christian P, West K Jr. Analyzing the mobile "digital divide": changing determinants of household phone ownership over time in rural bangladesh. JMIR Mhealth Uhealth. 2015 Feb 25;3(1):e24. doi: 10.2196/mhealth.3663. PMID 25720457
- [Derived] Tong H, Thorne-Lyman A, Palmer AC, Shaikh S, Ali H, Gao Y, Pasqualino MM, Wu L, Alland K, Schulze K, West KP Jr, Hossain MI, Labrique AB. Prelacteal feeding is not associated with infant size at 3 months in rural Bangladesh: a prospective cohort study. Int Breastfeed J. 2024 Feb 27;19(1):15. doi: 10.1186/s13006-024-00621-4. PMID 38413997